CLINICAL TRIAL: NCT06193824
Title: Characterization of the Endocrine Response to Exercise: Impact of the Muscle Contraction Modality
Brief Title: Optimisation of Eccentric Exercises
Acronym: OPTIMEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RBHP 2022 RANNOU
Record Dates: First submitted 2023-06-23; First posted 2024-01-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy Control Subjects

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- downhill treadmill walking -10% gradient (Experimental): The subjects will perform downhill walking at 6 km/h for 45 min on a treadmill (-10% incline)
  Interventions: Device: Experimental: downhill treadmill walking at -10% and -20% gradient
- downhill treadmill walking -20% gradient (Experimental): The subjects will perform downhill walking at 6 km/h for 45 min on a treadmill (-20% incline)
  Interventions: Device: Experimental: downhill treadmill walking at -10% and -20% gradient

INTERVENTIONS:
Device: Experimental: downhill treadmill walking at -10% and -20% gradient — The subjects will perform downhill walking at 6 km/h for 45 min on a treadmill (-10% or -20% incline)

SUMMARY:
Regular physical activity is an important public health lever and is recognised as an alternative in the management of certain long-term conditions. To achieve beneficial effects on the body, exercise recommendations are based on several parameters such as duration, intensity and continuous or intermittent nature of the activity. However, the mode of muscle contraction during exercise is generally little considered or poorly defined in these recommendations, which can lead to prescribing errors. In particular, the eccentric contraction modality, which can be found in actions designed to slow down movement (e.g. walking downhill), represents an interesting strategy, but its prescription modalities are still poorly understood.

The beneficial effects of physical activity are based in part on the release of molecules (myokines) by the skeletal muscles during exercise, which improve the functioning of the body. However, the effect of downhill walking on the release of myokines by the muscle has been little studied. The lack of knowledge of this effect is therefore an obstacle to the use of this exercise modality to try to optimise physical activity recommendations for health or performance improvement.

The aim of this study is therefore to better understand how downhill walking (eccentric muscle contraction) affects the production of molecules by muscles (myokines) during exercise.

DETAILED DESCRIPTION:
After being informed of the aims, nature and possible risks of the study, written informed consent will be obtained from the subjects.

Prior to enrolment, volunteers will undergo a medical evaluation that includes a review of personal and family medical history, any current medications, and a standard physical examination. Compliance with the inclusion/exclusion criteria will be checked during this examination.

After enrolment, subjects will perform a treadmill familiarization session.

Experimental days:

* Subjects will complete a 45-minute walking exercise on a negative gradient treadmill (6 km/h) in a randomised 2-way cross-over design with either a -10% or -20% gradient.
* Blood will be sampled immediately pre-exercise, 1-h and 24-h post-exercise for the analysis of muscle myokines.
* Exercise-induced muscle fatigue in lower limbs will be evaluated using squat and counter-movement jumps immediately before and post-exercise.
* Heart-rate variability will be measured during the eccentric exercise session.
* Thigh muscle volume will be measured immediately before and post-exercise.
* Exercise-induced myalgia at 24-, 48-, 72- and 96h will be assessed using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 24.9 kg/m² (18.5 ≤ BMI ≤ 24.9)
* Non-smoker
* No treatment (background or at the time of the examination)
* Physical check up considered compatible with study participation (no bones, articular or muscular problems in lower limbs)
* Subjects considered healthy by investigator based on medical questioning and clinical examination
* Affiliation to the French Social Security system
* Person who has read and understood the research-related information, and signed the consent forms

Exclusion Criteria:

* Smoking
* Subjects with heart or respiratory failure
* Participants with lower extremity injury in the past three months
* Contraindication to the application of a magnetic field (wearing a pacemaker, presence of prosthetic material or ferromagnetic foreign bodies, presence of cochlear implants or ocular prosthetic material)
* Participant that does not wish to participate (refusal to sign the consent form)
* Patients under guardianship, trusteeship, deprived of liberty or safeguard of justice

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effect of eccentric exercise on myokine concentrations | Blood sample at baseline (prior exercise), Hour 1 and Hour 24 post-exercise
  Changes in systemic myokine levels following submaximal downhill treadmill exercise at different inclines, at the same speed and for the same duration.
Effect of treadmill inclination on myokine concentrations | Blood sample at baseline (prior exercise), Hour 1 and Hour 24 post-exercise
  Differences in systemic myokine levels concentrations following -10 and -20% gradient submaximal downhill treadmill exercises, at the same speed and for the same duration.

SECONDARY OUTCOMES:
Assessment of exercise-induced muscle fatigue in lower limbs | Baseline (prior exercise) and 15 seconds post-exercise
  squat jump
Assessment of exercise-induced muscle fatigue in lower limbs | Baseline (prior exercise) and 15 seconds post-exercise
  counter-movement jump
Assessment of autonomic nervous system function | During treadmill exercise
  Heart rate variability (HRV) analysis Temporal and spectral analyses of cardiac variability
Effect of treadmill exercise on muscle volume | Baseline (prior exercise) and 15 seconds post-exercise
  Measurement of thigh and calf circumferences
Effect of treadmill exercise on muscle pain | Baseline (prior exercise) and 15 seconds post-exercise
  Measurement of muscle pain induced by a half-squat movement (self-measurement by the subject using a visual analogic scale, 0-10)
Effect of treadmill exercise on delayed onset muscle soreness | Baseline (prior exercise) and Hour 24, Hour 48, Hour 72, Hour 96 post-exercise
  Measurement of muscle pain induced by eccentric exercise (self-measurement by the subject using a visual analogic scale, 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France